CLINICAL TRIAL: NCT07371910
Title: A Randomized, Open-label, Controlled, Multicenter Phase III Study of Fluorizoparib in Combination With Apatinib Versus Investigator's Choice Chemotherapy in Patients With HRD-positive, HER2-negative Advanced Breast Cancer
Brief Title: Fluorizoparib Plus Apatinib Versus Chemotherapy in HRD-positive, HER2-negative Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1016-05
Record Dates: First submitted 2026-01-14; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer; HRD-Positive/HER2-Negative Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential Fluorizoparib + Apatinib after Chemotherapy/ADC (Experimental): This is the experimental arm. Participants receive a two-phase sequential treatment strategy:
  Induction Phase: 6 cycles of investigator-selected chemotherapy or ADC therapy.
  Maintenance Phase: Participants who complete induction without disease progression switch to long-term oral maintenance therapy with the combination of Fluorizoparib and Apatinib.
  Treatment continues until disease progression, unacceptable toxicity, withdrawal, or death.
  Interventions: Drug: Chemotherapy/ADC Regimen; Drug: Fluorizoparib; Drug: Apatinib
- Physician's Choice Chemotherapy/ADC Regimen (Active Comparator): This is the control arm intervention. Participants receive continuous treatment with a standard chemotherapy regimen or an Antibody-Drug Conjugate (ADC) selected by the investigator from protocol-specified options (e.g., eribulin, vinorelbine, gemcitabine, capecitabine, sacituzumab govitecan, or trastuzumab deruxtecan). Treatment is administered intravenously or orally according to the standard schedule of the chosen agent and continues without a planned switch to the oral targeted combination therapy, until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Interventions: Drug: Physician's Choice Chemotherapy/ADC Regimen

INTERVENTIONS:
Drug: Chemotherapy/ADC Regimen — This is the initial induction phase of the experimental arm. Participants will receive 6 cycles of a standard intravenous or oral chemotherapy regimen or an Antibody-Drug Conjugate (ADC), selected by the investigator from protocol-specified options (e.g., eribulin, vinorelbine, gemcitabine, capecitabine, sacituzumab govitecan, or trastuzumab deruxtecan). Administration follows the standard schedule of the chosen agent. The purpose is to achieve disease control before switching to long-term maintenance therapy.
  Arms: Sequential Fluorizoparib + Apatinib after Chemotherapy/ADC
Drug: Fluorizoparib — This oral PARP inhibitor is administered as part of the maintenance phase. Participants who complete the 6-cycle induction phase without disease progression switch to Fluorizoparib twice daily in continuous 21-day cycles, in combination with Apatinib, until disease progression or unacceptable toxicity.
  Arms: Sequential Fluorizoparib + Apatinib after Chemotherapy/ADC
Drug: Apatinib — This oral anti-angiogenic TKI is administered as part of the maintenance phase. Participants who complete the 6-cycle induction phase without disease progression switch to Apatinib once daily in continuous 21-day cycles, in combination with Fluorizoparib, until disease progression or unacceptable toxicity.
  Arms: Sequential Fluorizoparib + Apatinib after Chemotherapy/ADC
Drug: Physician's Choice Chemotherapy/ADC Regimen — Participants receive continuous treatment with a standard chemotherapy regimen or an Antibody-Drug Conjugate (ADC) selected by the investigator from protocol-specified options (e.g., eribulin, vinorelbine, gemcitabine, capecitabine, sacituzumab govitecan, or trastuzumab deruxtecan). Treatment is administered intravenously or orally according to the standard schedule of the chosen agent and continues without a planned switch to the oral targeted combination therapy, until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Arms: Physician's Choice Chemotherapy/ADC Regimen

SUMMARY:
This is a Phase III clinical trial for patients with a specific type of advanced breast cancer that is HER2-negative and has a biomarker called "Homologous Recombination Deficiency (HRD)-positive."

The study aims to compare the effectiveness and safety of two treatment strategies:

Experimental Group: Patients will first receive 6 cycles of standard chemotherapy or antibody-drug conjugate (ADC) therapy chosen by their doctor. After completing these 6 cycles, they will switch to a combination of two oral targeted drugs: Fluorizoparib and Apatinib, as long-term maintenance therapy.

Control Group: Patients will continue to receive their doctor's choice of standard chemotherapy or ADC therapy without switching to the targeted drug combination.

Patients will be randomly assigned (like flipping a coin) to one of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-70 years.

Histologically confirmed HER2-negative metastatic breast cancer.

Documented HRD-positive status (defined as BRCA1/2 mutation and/or HRD positive).

HR+/HER2- patients must have received prior endocrine therapy for metastatic disease.

Have received no more than 2 prior lines of chemotherapy or ADC therapy for metastatic disease.

At least one measurable lesion per RECIST 1.1.

ECOG performance status 0-2 and life expectancy ≥3 months.

Adequate organ function (bone marrow, liver, renal, cardiac).

Exclusion Criteria:

* HR+/HER2- patients who have not received prior endocrine therapy for metastatic disease.

Have not received any prior systemic therapy for metastatic breast cancer.

Have received >2 prior lines of chemotherapy or ADC therapy for metastatic disease.

Known severe hypersensitivity to any component of the study drugs.

Pregnant, lactating, or women of childbearing potential unwilling to use effective contraception.

Uncontrolled or significant cardiovascular disease.

Any other condition deemed inappropriate for the study by the investigato

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) | From randomization until disease progression or death (assessed up to approximately 4 years).
Progression-Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) | From randomization until disease progression or death (assessed up to approximately 4 years).
  The time from randomization to the first documented disease progression according to RECIST 1.1 criteria, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From randomization until first documented response or progression (assessed every 6-8 weeks during treatment, up to approximately 2 years)
Overall Survival (OS) | From randomization until death from any cause (assessed up to approximately 7 years, which is the total study duration)
Clinical Benefit Rate (CBR) | From randomization until progression or 24 weeks of stable disease (assessed up to approximately 2 years).
Disease Control Rate (DCR) | From randomization until the end of treatment or progression (assessed up to approximately 2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ray-Coquard I, Pautier P, Pignata S, Pérol D, González-Martín A, Berger R, Fujiwara K, Vergote I, Colombo N, Mäenpää J, Selle F, Sehouli J, Lorusso D, Guerra Alía EM,Reinthaller A, Nagao S, Lefeuvre-Plesse C, Canzler U, Scambia G, Lortholary A, Marmé F, Combe P, de Gregorio N, Rodrigues M, Buderath P, Dubot C, Burges A, You B, Pujade-Lauraine E, Harter P; PAOLA-1 Investigators. Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2416-2428.
- [Background] Liu JF, Barry WT, Birrer M, Lee JM, Buckanovich RJ, Fleming GF, Rimel B, Buss MK, Nattam S, Hurteau J, Luo W, Quy P, Whalen C, Obermayer L, Lee H, Winer EP, Kohn EC, Ivy SP, Matulonis UA. Combination cediranib and olaparib versus olaparib alone for women with recurrent platinum-sensitive ovarian cancer: a randomised phase 2 study. Lancet Oncol. 2014 Oct;15(11):1207-14.
- [Background] Liu JF, Barry WT, Birrer M, Lee JM, Buckanovich RJ, Fleming GF, Rimel BJ, Buss MK, Nattam SR, Hurteau J, Luo W, Curtis J, Whalen C, Kohn EC, Ivy SP, Matulonis UA. Overall survival and updated progression-free survival outcomes in a randomized phase II study of combination cediranib and olaparib versus olaparib in relapsed platinum-sensitive ovarian cancer. Ann Oncol. 2019 Apr 1;30(4):551-557.
- [Background] Gruber JJ, Afghahi A, Timms K, DeWees A, Gross W, Aushev VN, Wu HT, Balcioglu M, Sethi H, Scott D, Foran J, McMillan A, Ford JM, Telli ML. A phase II study of talazoparib monotherapy in patients with wild-type BRCA1 and BRCA2 with a mutation in other homologous recombination genes. Nat Cancer. 2022 Oct;3(10):1181-1191.
- [Background] Severson TM, Wolf DM, Yau C, Peeters J, Wehkam D, Schouten PC, Chin SF, Majewski IJ, Michaut M, Bosma A, Pereira B, Bismeijer T, Wessels L, Caldas C, Bernards R, Simon IM, Glas AM, Linn S, van 't Veer L. The BRCA1ness signature is associated significantly with response to PARP inhibitor treatment versus control in the I-SPY 2 randomized neoadjuvant setting. Breast Cancer Res. 2017 Aug 25;19(1):99.
- [Background] Sun C, Yin J, Fang Y, Chen J, Jeong KJ, Chen X, Vellano CP, Ju Z, Zhao W, Zhang D, Lu Y, Meric-Bernstam F, Yap TA, Hattersley M, O'Connor MJ, Chen H, Fawell S, Lin SY, Peng G, Mills GB. BRD4 Inhibition Is Synthetic Lethal with PARP Inhibitors through the Induction of Homologous Recombination Deficiency. Cancer Cell. 2018 Mar 12;33(3):401-416.e8.
- [Background] Ray-Coquard I, Pautier P, Pignata S, Pérol D, González-Martín A, Berger R, Fujiwara K, Vergote I, Colombo N, Mäenpää J, Selle F, Sehouli J, Lorusso D, Guerra Alía EM, Reinthaller A, Nagao S, Lefeuvre-Plesse C, Canzler U, Scambia G, Lortholary A, Marmé F, Combe P, de Gregorio N, Rodrigues M, Buderath P, Dubot C, Burges A, You B, Pujade-Lauraine E, Harter P; PAOLA-1 Investigators. Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2416-2428.
- [Background] González-Martín A, Pothuri B, Vergote I, DePont Christensen R, Graybill W, Mirza MR, McCormick C, Lorusso D, Hoskins P, Freyer G, Baumann K, Jardon K, Redondo A, Moore RG, Vulsteke C, O'Cearbhaill RE, Lund B, Backes F, Barretina-Ginesta P, Haggerty AF, Rubio-Pérez MJ, Shahin MS, Mangili G, Bradley WH, Bruchim I, Sun K, Malinowska IA, Li Y, Gupta D, Monk BJ; PRIMA/ENGOT-OV26/GOG-3012 Investigators. Niraparib in Patients with Newly Diagnosed Advanced Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2391-2402.
- [Background] Annals of Oncology (2020) 31 (suppl_4): S551-S589. 10.1016/annonc/annonc276
- [Background] Robson M, Im SA, Senkus E, Xu B, Domchek SM, Masuda N, Delaloge S, Li W, Tung N, Armstrong A, Wu W, Goessl C, Runswick S, Conte P. Olaparib for Metastatic Breast Cancer in Patients with a Germline BRCA Mutation. N Engl J Med. 2017 Aug 10;377(6):523-533
- [Background] Litton JK, Rugo HS, Ettl J, Hurvitz SA, Gonçalves A, Lee KH, Fehrenbacher L,Yerushalmi R, Mina LA, Martin M, Roché H, Im YH, Quek RGW, Markova D, Tudor IC,Hannah AL, Eiermann W, Blum JL. Talazoparib in Patients with Advanced Breast Cancer and a Germline BRCA Mutation. N Engl J Med. 2018 Aug 23;379(8):753-763.
- [Background] Iglehart JD, Silver DP. Synthetic lethality--a new direction in cancer-drug development. N Engl J Med. 2009 Jul 9;361(2):189-91.
- [Background] Litton JK, Rugo HS, Ettl J, Hurvitz SA, Gonçalves A, Lee KH, Fehrenbacher L, Yerushalmi R, Mina LA, Martin M, Roché H, Im YH, Quek RGW, Markova D, Tudor IC, Hannah AL, Eiermann W, Blum JL. Talazoparib in Patients with Advanced Breast Cancer and a Germline BRCA Mutation. N Engl J Med. 2018 Aug 23;379(8):753-763.